CLINICAL TRIAL: NCT06260163
Title: A Phase 3 Randomized, Open-label Induction, Double-blind Maintenance, Parallel-group, Multicenter Protocol to Evaluate the Efficacy, Safety, and Pharmacokinetics of Guselkumab in Pediatric Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Guselkumab in Pediatric Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: QUASAR Jr
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109251; CNTO1959PUC3001 (Other: Janssen Research & Development, LLC); 2022-001285-35 (EudraCT Number); 2022-502238-22-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Open-label Induction Phase: Guselkumab Intravenously (IV) (Experimental): Participants will receive a guselkumab dose IV based on their body weight (BW) during the 12-week open-label induction phase.
  Interventions: Drug: Guselkumab Intravenous
- Open-label Induction Phase: Guselkumab Subcutaneously (SC) (Experimental): Participants will receive a guselkumab dose SC based on their BW during the 12-week open-label induction phase.
  Interventions: Drug: Guselkumab Subcutaneous
- Double-blind Maintenance Phase: Guselkumab Dose Regimen 1 (Experimental): At the end of the induction phase, Week 12 responders will be randomized into the double-blind maintenance phase to receive guselkumab dose regimen 1 SC based on their BW up to Week 56.
  Interventions: Drug: Guselkumab Subcutaneous
- Double-blind Maintenance Phase: Guselkumab Dose Regimen 2 (Experimental): At the end of the induction phase, Week 12 responders will be randomized into the double-blind maintenance phase to receive guselkumab dose regimen 2 SC based on their BW up to Week 56.
  Interventions: Drug: Guselkumab Subcutaneous
- Open-label Maintenance Phase: Guselkumab SC (Experimental): Week 12 non-responders will not be randomized and will enter an open-label maintenance phase to receive guselkumab SC dosing regimen based on their body weight up to Week 56.
  Interventions: Drug: Guselkumab Subcutaneous

INTERVENTIONS:
Drug: Guselkumab Subcutaneous — Guselkumab will be administered subcutaneously.
  Other Names: CNTO1959; TREMFYA
  Arms: Double-blind Maintenance Phase: Guselkumab Dose Regimen 1; Double-blind Maintenance Phase: Guselkumab Dose Regimen 2; Open-label Induction Phase: Guselkumab Subcutaneously (SC); Open-label Maintenance Phase: Guselkumab SC
Drug: Guselkumab Intravenous — Guselkumab will be administered intravenously.
  Other Names: CNTO1959; TREMFYA
  Arms: Open-label Induction Phase: Guselkumab Intravenously (IV)

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab in pediatric participants with moderately to severely active ulcerative colitis at the end of maintenance therapy among participants who were induction responders.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than or equal to (>=) 10 kilogram (kg) at the time of consent for screening
* A pathology report to support a documented diagnosis of Ulcerative Colitis (UC) must be available in the source documents. There is no maximum duration for which a participant needs to be diagnosed with UC. If the pathology report to support a documented diagnosis of UC is not available in the source documents, the screening endoscopy with biopsies (obtained within 3 weeks before first study intervention administration) needs to support the diagnosis of UC.
* Moderately to severely active UC, defined by a baseline modified Mayo (without physician's global assessment) score of 5 through 9 inclusive, with a screening Mayo endoscopy subscore >= 2 as determined by a central review of the video of the endoscopy
* Medically stable based on physical examination, medical history, and vital signs, performed at screening. Any abnormalities must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and acknowledged by the investigator
* Participants must have had an inadequate response and/or intolerance to biologic therapy and/or conventional therapies or be dependent upon corticosteroids

Exclusion Criteria:

* Have UC limited to the rectum only or to less than (<) 20 centimeter of the colon
* Presence of a stoma
* Has had any kind of bowel resection within 6 months or any other intra-abdominal surgery within 3 months of baseline
* Have severe colitis or have evidence of Crohn's Disease (CD)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2028-05-22 (Estimated); Study Completion 2028-08-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 56 | Week 56
  Percentage of participants with clinical remission as assessed by modified Mayo score at Week 56 among participants who were induction responders will be reported. Clinical remission per modified Mayo score is defined as a stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Response at Week 12 | Week 12
  Percentage of participants with clinical response as assessed by modified Mayo score at Week 12 will be reported. Modified Mayo score is a 3-component (stool frequency, rectal bleeding, and endoscopy subscores) assessment and does not include the physician's global assessment. A decrease from baseline in the modified Mayo score by greater than or equal to (>=) 30 percent and >= 2 points, with either a decrease from baseline in the rectal bleeding subscore of >= 1 or a rectal bleeding subscore of 0 or 1.
Percentage of Participants with Clinical Remission at Week 12 | Week 12
  Percentage of participants with clinical remission at Week 12 as assessed by modified Mayo score will be reported. Clinical remission per modified Mayo score is defined as a stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline.
Percentage of Participants With Pediatric Ulcerative Colitis Activity Index (PUCAI) Remission at Week 12 | Week 12
  Percentage of participants with PUCAI remission at Week 12 will be reported. It comprises 6 scales and ranges between 0 and 85 points. The scales are abdominal pain, rectal bleeding, stool consistency, number of stools, nocturnal bowel movement, and activity level. The PUCAI score is calculated as the sum of the 6 subscores. A PUCAI score of less than (<) 10 indicates remission.
Percentage of Participants with Symptomatic Remission at Week 12 | Week 12
  Percentage of participants with symptomatic remission at Week 12 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0, where the stool frequency subscore has not increased from induction baseline.
United States: Percentage of Participants with Endoscopic Improvement at Week 12 | Week 12
  Percentage of participants with endoscopic improvement as assessed by Mayo endoscopy subscore at Week 12 will be reported. Endoscopic improvement is defined as the Mayo endoscopy subscore of 0 or 1 with no friability present on the endoscopy.
European Union: Percentage of Participants with Endoscopic Healing at Week 12 | Week 12
  Percentage of participants with endoscopic healing as assessed by Mayo endoscopy subscore at Week 12 will be reported. Endoscopic healing is defined as the Mayo endoscopy subscore of 0 or 1 with no friability present on the endoscopy.
Percentage of Participants with Clinical Response at Week 56 | Week 56
  Percentage of participants with clinical response as assessed by modified Mayo score at Week 56 will be reported. Modified Mayo score is a 3-component (stool frequency, rectal bleeding, and endoscopy subscores) assessment and does not include the physician's global assessment. A decrease from baseline in the modified Mayo score by >= 30 percent and >= 2 points, with either a decrease from baseline in the rectal bleeding subscore of >= 1 or a rectal bleeding subscore of 0 or 1.
Percentage of Participants With PUCAI Remission at Week 56 | Week 56
  Percentage of participants with PUCAI remission at Week 56 will be reported. PUCAI comprises of 6 scales and ranges between 0 and 85 points. The scales are: abdominal pain, rectal bleeding, stool consistency, number of stools, nocturnal bowel movement, and activity level. The PUCAI score is calculated as the sum of the 6 subscores. A PUCAI score of less than (<) 10 indicates remission.
Percentage of Participants with Symptomatic Remission at Week 56 | Week 56
  Percentage of participants with symptomatic remission at Week 56 will be reported. Symptomatic remission is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0, where the stool frequency subscore has not increased from induction baseline.
Percentage of Participants with Symptomatic Remission at Week 56 Among Participants who had Symptomatic Remission at Week 12 | Week 56
  Percentage of participants with symptomatic remission at Week 56 among participants who had symptomatic remission at Week 12 will be reported. Symptomatic remission score is defined as a stool frequency subscore of 0 or 1 and a rectal bleeding subscore of 0, where the stool frequency subscore has not increased from induction baseline.
United States: Percentage of Participants With Endoscopic Improvement at Week 56 | Week 56
  Percentage of participants with endoscopic improvement as assessed by Mayo endoscopy subscore at Week 56 will be reported. Endoscopic improvement is defined as the Mayo endoscopy subscore of 0 or 1 with no friability present on the endoscopy.
European Union: Percentage of Participants With Endoscopic Healing at Week 56 | Week 56
  Percentage of participants with endoscopic healing as assessed by Mayo endoscopy subscore at Week 56 will be reported. Endoscopic healing is defined as the Mayo endoscopy subscore of 0 or 1 with no friability present on the endoscopy.
Percentage of Participants Who Achieve Endoscopic Normalization at Week 56 | Week 56
  Percentage of participants who achieve endoscopic normalization with an endoscopy subscore of 0 at Week 56 will be reported.
Percentage of Participants Histo-endoscopic Mucosal Improvement at Week 56 | Week 56
  Percentage of participants histo-endoscopic mucosal healing per endoscopy subscore and histologic improvement at Week 56 will be reported. Histologic-endoscopic mucosal healing is defined as achieving a combination of histologic improvement and endoscopic improvement (US) or endoscopic healing (EU) (endoscopy subscore of 0 or 1).
Percentage of Participants with Corticosteroid-free Clinical Remission at Week 56 | Week 56
  Percentage of participants with corticosteroid-free clinical remission at Week 56 will be reported. Corticosteroid free clinical remission is defined as a Mayo stool frequency subscore of 0 or 1, a rectal bleeding subscore of 0, and an endoscopy subscore of 0 or 1 with no friability present on the endoscopy, where the stool frequency subscore has not increased from induction baseline (Week 0), and not receiving corticosteroids for at least 8 weeks prior to Week 56
Serum Concentration of Guselkumab During Induction Phase | From Week 0 to Week 12
  Serum samples will be analyzed to determine concentrations of guselkumab overtime.
Serum Concentration of Guselkumab During Maintenance Phase | From Week 12 to Week 56
  Serum samples will be analyzed to determine concentrations of guselkumab over time.
Number of Participants with Incidence of Anti-guselkumab Antibodies | Up to Week 68
  Number of participants with anti-guselkumab antibodies for all study treatment regimens will be assessed.
Percentage of Participants with Adverse Events (AEs) | Up to Week 68
  Percentage of participants with AEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 68
  Percentage of participants with SAEs will be reported. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly.
Percentage of Participants with AEs Leading to Discontinuation of Study Intervention | Up to Week 68
  Percentage of participants with AEs leading to discontinuation of study intervention will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (61):
- United States (3):
  - Children's Hospital Oakland, Oakland, California
  - Riley Hospital for Children, Indianapolis, Indiana
  - NYU Langone Health, Lake Success, New York
- Australia (3):
  - The Kids Research Institute Australia on behalf of the Centre for Child Health Research, Nedlands
  - Mater Hospital Brisbane Inflammatory Bowel Diseases, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Belgium (4):
  - CHU Charleroi Chimay, Charleroi
  - UZ Gent, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
- China (8):
  - Capital Center For Children's health Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Changzhou No 2 Peoples Hospital, Changzhou
  - The Childrens Hospital Zhejiang University School Of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Henan Children's Hospital, Zhengzhou Children's Hospital, Zhengzhou
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N
  - Hvidovre Hospital, Hvidovre
- France (5):
  - Hospices Civils de Lyon - Groupement Hospitalier Est - Hopital Femme Mere Enfant, Bron
  - Hopital Francois Mitterand, Dijon
  - CHRU Lille, Lille
  - APHP Hopital Robert Debre, Paris
  - CHU Toulouse, Toulouse
- Italy (8):
  - ASST Papa Giovanni XXIII Bergamo, Bergamo
  - Azienda USL di Bologna - Ospedale Maggiore, Bologna
  - AOU Meyer, Florence
  - Ospedale S. Spirito, Azienda Sanitaria Pescara, Pescara
  - AOU Policlinico Umberto I, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - IRCCS Materno Infantile Burlo Garofolo, Trieste
- Japan (10):
  - Tokyo Metropolitan Children's Medical Center, Fuchū
  - Kanazawa University Hospital, Kanazawa
  - Kobe University Hospital, Kobe
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Shinshu University Hospital, Matsumoto
  - Saga University Hospital, Saga
  - National Center for Child Health and Development, Setagaya Ku
  - Tokyo Medical University Hospital, Shinjuku
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama
- Norway (4):
  - Akershus Universitetssykehus, Lørenskog
  - Oslo University Hospital, Oslo
  - Universitetssykehuset Nord-Norge HF, Tromsø
  - St. Olavs Hospital, Trondheim
- Poland (4):
  - Copernicus Podmiot Leczniczy Sp. z o.o, Gdansk
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - Medical Network Spolka z o.o. WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Portugal (3):
  - Uls Santa Maria - Hosp. Santa Maria, Lisbon
  - Uls Santo Antonio - Cmin, Porto
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- Spain (3):
  - Hosp. Infantil Univ. Nino Jesus, Madrid
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. I Politecni La Fe, Valencia
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Marmara University Pendik Training Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency